CLINICAL TRIAL: NCT06557902
Title: An Open-label, Multiple-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Lumateperone in Pediatric Patients, Ages 5 to Less Than 13 Years, Diagnosed With Autism Spectrum Disorder
Brief Title: Safety, Tolerability and Pharmacokinetics of Lumateperone in Pediatric Patients With Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-035
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — lumateperone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (10 to less than 13 years) (Experimental): Lumateperone capsule once daily: 10.5 mg on Days 1 and 2; 10.5 mg or 21 mg on Day 3; 10.5 mg or 21 mg on Days 4 and 5
  Interventions: Drug: Lumateperone 10.5 mg capsule; Drug: Lumateperone 21 mg capsule
- Group 2 (5 to less than 10 years) (Experimental): Lumateperone ODT once daily: 5 mg on Days 1 and 2; 5 mg or 10.5 mg on Day 3; 5 mg or 10.5 mg on Days 4 and 5; dosing regimen may be adjusted after the first 6 patients dosed and will not exceed 21 mg in subsequent patients
  Interventions: Drug: Lumateperone 5 mg ODT; Drug: Lumateperone 10.5 mg ODT; Drug: Lumateperone 15.5 mg ODT; Drug: Lumateperone 21 mg ODT

INTERVENTIONS:
Drug: Lumateperone 10.5 mg capsule — Lumateperone 10.5 mg capsule, oral administration
  Arms: Group 1 (10 to less than 13 years)
Drug: Lumateperone 21 mg capsule — Lumateperone 21 mg capsule, oral administration
  Arms: Group 1 (10 to less than 13 years)
Drug: Lumateperone 5 mg ODT — Lumateperone 5 mg ODT, oral administration
  Arms: Group 2 (5 to less than 10 years)
Drug: Lumateperone 10.5 mg ODT — Lumateperone 10.5 mg ODT, oral administration
  Arms: Group 2 (5 to less than 10 years)
Drug: Lumateperone 15.5 mg ODT — Lumateperone 5 mg ODT + 10.5 mg ODT, oral administration
  Arms: Group 2 (5 to less than 10 years)
Drug: Lumateperone 21 mg ODT — Lumateperone 21 mg ODT, oral administration
  Arms: Group 2 (5 to less than 10 years)

SUMMARY:
Study ITI-007-035 is a Phase 1b, multicenter, open-label study to evaluate the safety, tolerability, and PK of lumateperone for pediatric patients with Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 5 to less than 13 years of age
* Primary clinical diagnosis of ASD with symptoms of irritability
* ABC-I subscale score of ≥12 at Screening
* CGI-S score of ≥3 at Screening
* Body mass index (BMI) greater than the 5th percentile according to age- and gender-specific CDC Clinical Growth Charts (2000) at Screening
* Ability to swallow capsules

Exclusion Criteria:

* Has a primary psychiatric diagnosis other than ASD
* Reports suicidal ideation (Type 3, 4 or 5 on the Baseline/Screening version of the C-SSRS) within 6 months prior to Screening, or any suicidal behavior within 2 years prior to Screening, and/or the Investigator assesses the patient to be a safety risk to him/herself or others
* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the patient at risk or interfere with study outcome variables
* History of a clinically significant cardiac disorder and/or abnormal screening ECG or a QT interval corrected for heart rate using Fridericia formula (QTcF) > 460 msec at Screening
* Patients with a history of orthostatic hypotension or who have orthostatic hypotension at Screening
* Has a history of uncontrolled/disruptive behavior in the past 30 days that, in the Investigator's opinion, would preclude the ability to participate in study procedures

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Cmax | Day 5
  Maximum plasma concentration of lumateperone
Pharmacokinetics: Tmax | Day 5
  Time of maximum plasma concentration of lumateperone
Pharmacokinetics: AUC0-tau | Day 5
  Area under the plasma lumateperone concentration time curve from time zero to the end of dosing (tau)

SECONDARY OUTCOMES:
Percentage of patients with treatment-emergent adverse events | Up to 30 days after last dose
Change from baseline in systolic and diastolic blood presssure | Day 6
Change from baseline in ECG QT interval | Day 6
Change from baseline in hemoglobin | Day 6
Change from baseline in white blood cell count | Day 6
Change from baseline in aspartate aminotransferase | Day 6
Change from baseline in alanine aminotransferase | Day 6
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | Day 6
  AIMS is a measure of facial and oral movements, extremity movements and trunk movements. Items are rated on a scale from none (0) to severe (4).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Clinical Site 6, Miami, Florida
  - Clinical Site 7, Orlando, Florida
  - Clinical Site 1, Atlanta, Georgia
  - Clinical Site 2, Decatur, Georgia
  - Clinical Site 3, Savannah, Georgia
  - Clinical Site 4, Saint Charles, Missouri
  - Clinical Site 5, Lincoln, Nebraska
  - Clinical Site 8, Everett, Washington

IPD SHARING:
Plan to Share IPD: No